CLINICAL TRIAL: NCT00723710
Title: Guidelines to the Intron A® Health Management Program II: A Nursing Support Program for Patients With High-Risk Melanoma Receiving High Dose Intron A Therapy
Brief Title: Effect of Proactive Management of Side Effects on Treatment Compliance in Malignant Melanoma Patients on High-dose Intron A Therapy (Study P04600)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04600
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2013-10-28 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Introns; Interferon alpha-2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intron A: Patients with malignant melanoma who are free of disease post-surgery but at high risk for systemic recurrence.
  Interventions: Biological: Intron A (interferon alfa-2b; SCH 30500)

INTERVENTIONS:
Biological: Intron A (interferon alfa-2b; SCH 30500) — The recommended regimen includes an induction treatment of 5 consecutive days per week for 4 weeks as a 20-minute intravenous (iv) infusion at a dose of 20 million international units per square meter (MIU/m^2). The induction treatment should be followed by a maintenance treatment of 3 times per week for 48 weeks as a subcutaneous (sc) injection at a dose of 10 MIU/m^2. Therapy should be administered for a total of one year unless the disease progresses or the treatment has lead to recurrent unmanageable serious adverse effects.
  Other Names: SCH 30500

SUMMARY:
Patients with malignant melanoma who had undergone surgery will receive adjuvant treatment with high-dose Intron A for one year. The objective of this study is to maximize treatment compliance by proactive management of side effects in a day-to-day healthcare setting.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age > 18 years
* Confirmed melanoma
* Patient has been prescribed Intron A therapy for High-Risk Stage II & III Melanoma
* Intron A therapy started within 70 days of surgery (additional 15 days may be granted by the sponsor upon written approval)
* Proper contraception in both male and female subjects and the female partner(s) of male study subjects

Exclusion Criteria:

* Metastatic disease at the time of diagnosis
* Other malignancies
* History of non compliance to other therapies
* Pregnancy or breast feeding
* Previous Intron A therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 300 patients with malignant melanoma who are free of disease but at high risk for systemic recurrence. The study is conducted in Canada.
Sampling Method: Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2006-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

REFERENCES:
- [Result] Levesque N, Mitchinson K, Lawrie D, Fedorak L, Macdonald D, Normand C, Pouliot JF. Health management program: factors influencing completion of therapy with high-dose interferon alfa-2b for high-risk melanoma. Curr Oncol. 2008 Jan;15(1):36-41. doi: 10.3747/co.2008.200. PMID 18317583

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 299 participants were enrolled. Of these, 294 were considered efficacy evaluable (5 participants were excluded from efficacy analyses: 2 moved, 1 required radiation, 1 not eligible and 1 missing data).
Groups:
- Intron A: The recommended regimen included an induction treatment of 5 consecutive days per week for 4 weeks as a 20-minute intravenous (iv) infusion at a dose of 20 million international units per square meter (MIU/m^2). The induction treatment was followed by a maintenance treatment of 3 times per week for 48 weeks as a subcutaneous (sc) injection at a dose of 10 MIU/m^2. Therapy was administered for a total of one year unless the disease progressed or the treatment led to recurrent unmanageable serious adverse effects.
Period: Overall Study
Arm/Group | Intron A
Started | 294
Completed | 120
Not Completed | 174
Not completed — Disease progression | 48
Not completed — Adverse Event | 88
Not completed — Withdrawal by Subject | 36
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Groups:
- Intron A: The recommended regimen included an induction treatment of 5 consecutive days per week for 4 weeks as a 20-minute intravenous (iv) infusion at a dose of 20 MIU/m^2. The induction treatment was followed by a maintenance treatment of 3 times per week for 48 weeks as a subcutaneous (sc) injection at a dose of 10 MIU/m^2. Therapy was administered for a total of one year unless the disease progressed or the treatment led to recurrent unmanageable serious adverse effects.
Arm/Group | Intron A
Number analyzed (Participants) | 294
Age, Continuous [Median (Full Range); unit: years] | 52 [19 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124
  Male | 170

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Treatment
Description: Treatment completion was defined as those who completed both the induction and maintenance phases.
Time Frame: Up to 1 year
Population: The number of participants who started the induction phase
Measure: Number; unit: Participants
Arm/Group | Intron A
Number analyzed (Participants) | 294
Participants | 120

ADVERSE EVENTS:
Description: Population was all enrolled participants (299).
Arm/Group | Intron-A
Serious Adverse Events (participants affected / at risk) | 21/299
Other Adverse Events (participants affected / at risk) | 297/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intron-A (N=299)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
VISUAL IMPAIRMENT (Eye disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 2 (2)
CHILLS (General disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
INFUSION SITE SWELLING (General disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1)
CELLULITIS (Infections and infestations) | 2 (2)
GROIN ABSCESS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1)
SEROMA (Injury, poisoning and procedural complications) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
PRIMARY SEQUESTRUM (Musculoskeletal and connective tissue disorders) | 1 (1)
FEMALE REPRODUCTIVE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
DIZZINESS (Nervous system disorders) | 1 (1)
GRAND MAL CONVULSION (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 3 (3)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
OBSESSIVE-COMPULSIVE DISORDER (Psychiatric disorders) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1)
THROAT TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intron-A (N=299)
NEUTROPENIA (Blood and lymphatic system disorders) | 69 (114)
CONSTIPATION (Gastrointestinal disorders) | 32 (37)
DIARRHOEA (Gastrointestinal disorders) | 60 (81)
DRY MOUTH (Gastrointestinal disorders) | 18 (21)
DYSPEPSIA (Gastrointestinal disorders) | 18 (19)
NAUSEA (Gastrointestinal disorders) | 159 (224)
VOMITING (Gastrointestinal disorders) | 68 (88)
ASTHENIA (General disorders) | 17 (23)
CHILLS (General disorders) | 35 (56)
FATIGUE (General disorders) | 189 (275)
INFLUENZA LIKE ILLNESS (General disorders) | 220 (256)
PYREXIA (General disorders) | 86 (103)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 117 (155)
WEIGHT DECREASED (Investigations) | 26 (29)
DECREASED APPETITE (Metabolism and nutrition disorders) | 80 (105)
MYALGIA (Musculoskeletal and connective tissue disorders) | 84 (102)
DIZZINESS (Nervous system disorders) | 18 (24)
DYSGEUSIA (Nervous system disorders) | 50 (60)
HEADACHE (Nervous system disorders) | 145 (215)
ANXIETY (Psychiatric disorders) | 20 (22)
DEPRESSION (Psychiatric disorders) | 97 (102)
INSOMNIA (Psychiatric disorders) | 28 (36)
COUGH (Respiratory, thoracic and mediastinal disorders) | 33 (41)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 21 (22)
ALOPECIA (Skin and subcutaneous tissue disorders) | 29 (29)
PRURITUS (Skin and subcutaneous tissue disorders) | 19 (20)
RASH (Skin and subcutaneous tissue disorders) | 36 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No